CLINICAL TRIAL: NCT01368432
Title: Escitalopram (Lexapro) for the Treatment of TBI Depression and Other Comorbid Psychiatric Conditions
Brief Title: Lexapro for the Treatment of Traumatic Brain Injury (TBI) Depression & Other Psychiatric Conditions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Vani Rao, MD, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00020154
Record Dates: First submitted 2011-06-03; First posted 2011-06-08 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: TBI; Major Depression; Other Psychiatric Disorders
Keywords: TBI; Depression; Mood; Behavior
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Behavior | interventions — Escitalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Daily for 12 weeks
  Interventions: Drug: Placebo
- Escitalopram (Experimental): Escitalopram 10 mg or 20 mg daily for 12 weeks
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10 mg or 20 mg daily for 12 weeks by mouth
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — Sugar pill placebo
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This research is being done to see if a drug called escitalopram (Lexapro) is helpful to people who are suffering from depression after traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Despite it's high prevalence, little is known about the pharmacological treatment of depression following Traumatic Brain Injury (TBI). This is because of a lack of randomized controlled studies in the treatment of post-TBI depression. This study is designed to examine the safety and effectiveness of escitalopram in the treatment of post-TBI depression. It will also investigate metabolic changes and neural pathways associated with post-TBI depression and metabolic alterations after treatment through neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Closed head injury
* Fulfill Diagnostic and Statistical Manual Diploma in Social Medicine (DSM) IV criteria "Major Depressive Disorder"
* 18 years of age or older
* Able to provide informed consent
* Stable medical history

Exclusion Criteria:

* History of Stroke, Encephalitis, Seizures, or any other pre-TBI neurological diseases
* History of mental retardation
* Alcohol or Substance dependence in the last 1 year
* Inability to undergo MRI scan
* Pregnancy
* Current use of any psychotropic medications including any antidepressants, antipsychotics, anxiolytics, or sedative hypnotics
* Poor response to escitalopram in the past
* Acutely suicidal or requiring inpatient psychiatric hospitalization, as determined by the study psychiatrist
* Good medication response to another antidepressant in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vani Rao, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Brain Injury Association of Maryland — http://www.biamd.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Brain injury clinic at Johns Hopkins Bayview Medical Center, other Johns Hopkins outpatient clinics, and via advertisements in local papers.
Pre-assignment Details: One admitted to active alcohol abuse before initiating medications , and therefore no longer met inclusion criteria. Another consented but failed to return for any follow-up visits.
Groups:
- Placebo: The placebo group received a pill which appeared similar to the 10 and 20 mg of escitalopram.
- Escitalopram: Escitalopram was started at 10 mg per day and increased to 20 mg if deemed clinically necessary, at week 4. No medication changes were made after week 8.
Period: Overall Study
Arm/Group | Placebo | Escitalopram
Started | 6 | 8
Completed | 6 | 7
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Escitalopram | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) at Baseline
Description: This scale assesses the range of symptoms most frequently observed in patients with major depression. This measure will be used to assess the difference in Montgomery-Asberg Depression Rating Scale (MADRS) at baseline and 12 weeks. The scores range from 0-60.
  0 to 6 - normal; 7 to 19 - mild depression; 20 to 34 - moderate depression; >34 - severe depression.
  In this study the score was used as a continuous variable.
Time Frame: MADRS score at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group Baseline: The placebo group received a pill which appeared similar to the 10 and 20 mg of escitalopram.
- Treatment Group Baseline: Escitalopram was started at 10 mg per day and increased to 20 mg if deemed clinically necessary, at week 4. No medication changes were made after week 8.
Arm/Group | Placebo Group Baseline | Treatment Group Baseline
Number analyzed (Participants) | 6 | 8
units on a scale | 29.5 (3.9) | 33.6 (6.9)

2. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 1
Time Frame: MADRS score at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group MADRS 12 Weeks: This group consists of participants who received the placebo intervention and their level of depression as assessed by the MADRS scoring system.
- Treatment Group MADRS 12 Weeks: This group consists of participants who received escitalopram and their level of depression as assessed by the MADRS scoring system.
Arm/Group | Placebo Group MADRS 12 Weeks | Treatment Group MADRS 12 Weeks
Number analyzed (Participants) | 6 | 8
units on a scale | 11.2 (9.5) | 7 (5.7)

3. Secondary Outcome: Clinical Global Impression (CGI) - Severity at Baseline
Description: This outcome measure is assessing the participant's overall psychiatric health based upon the CGI score as assessed by the investigator. Scores range from 1-7
  1. = Normal-not at all ill
  2. = Borderline mentally ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill patients.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group Baseline: This group consists of participants who received the placebo intervention and represents their baseline global health.
- Treatment Group Baseline: This group consists of participants who received escitalopram and represents their baseline global health
Arm/Group | Placebo Group Baseline | Treatment Group Baseline
Number analyzed (Participants) | 6 | 8
units on a scale | 4.5 (0.5) | 4.8 (0.5)

4. Secondary Outcome: Clinical Global Impression (CGI)- Improvement
Description: This outcome measure is assessing the participant's overall psychiatric health based upon the CGI score as assessed by the investigator.
  The scores range from 1-7
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
Time Frame: at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group 12 Weeks: This group consists of participants who received the placebo intervention and represents their global health score at 12 weeks
- Treatment Group 12 Weeks: This group consists of participants who received escitalopram and represents their global health at 12 weeks.
Arm/Group | Placebo Group 12 Weeks | Treatment Group 12 Weeks
Number analyzed (Participants) | 6 | 8
units on a scale | 2.7 (1.2) | 2.1 (0.6)

5. Secondary Outcome: Clinical Anxiety Scale (CAS)
Description: This outcome measure is assessing the participant's anxiety as assessed by the CAS.
  The scores range from 0( normal; no anxiety) to 21 ( severe anxiety). It is used as a continuous variable.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group Baseline: This group consists of participants who received the placebo intervention and represents their anxiety score.
- Treatment Group Baseline: This group consists of participants who received escitalopram intervention and represents their anxiety score.
Arm/Group | Placebo Group Baseline | Treatment Group Baseline
Number analyzed (Participants) | 6 | 8
units on a scale | 9.8 (3.8) | 14.8 (6.7)

6. Secondary Outcome: Clinical Anxiety Scale (CAS)
Description: as for outcome 5
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group 12 Weeks: This group consists of participants who received the placebo intervention and represents their anxiety score.
- Treatment Group 12 Weeks: This group consists of participants who received escitalopram intervention and represents their anxiety score.
Arm/Group | Placebo Group 12 Weeks | Treatment Group 12 Weeks
Number analyzed (Participants) | 6 | 8
units on a scale | 6.3 (4.3) | 3.9 (5)

7. Secondary Outcome: Satisfaction With Life (SWL)
Description: This outcome measure asses the participants overall satisfaction with life as measured by the SWL scale.
  The scores range from 5 ( absolutely no satisfaction ) to 35 ( very satisfied with life).
  It is used as continuous variable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group Baseline: This group consists of participants who received the placebo intervention.
- Treatment Group Baseline: This group consists of participants who received escitalopram intervention.
Arm/Group | Placebo Group Baseline | Treatment Group Baseline
Number analyzed (Participants) | 6 | 8
units on a scale | 13.8 (7.7) | 15.6 (9.3)

8. Secondary Outcome: Satisfaction With Life (SWL)
Description: as for outcome 7
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group 12 Weeks: This group consists of participants who received the placebo intervention.
- Treatment Group 12 Weeks: This group consists of participants who received escitalopram intervention.
Arm/Group | Placebo Group 12 Weeks | Treatment Group 12 Weeks
Number analyzed (Participants) | 6 | 8
units on a scale | 21.2 (9.2) | 22.6 (5.7)

9. Secondary Outcome: Quality of Life (QWL)
Description: This outcome measure is assessing the participants impression of their quality of life as measured by the QWL scale.
  Scores range from 16 ( terrible quality of life ) to 112 (Very delighted). Used as a continuous variable.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group Baseline | Treatment Group Baseline
Number analyzed (Participants) | 6 | 8
units on a scale | 62.8 (22.3) | 64.1 (24.6)

10. Secondary Outcome: Quality of Life (QWL)
Description: as for outcome 9
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group 12 Weeks | Treatment Group 12 Weeks
Number analyzed (Participants) | 6 | 8
units on a scale | 75.2 (30.3) | 78.7 (17.3)

11. Secondary Outcome: Disability Rating Scale (DRS)
Description: This scale is a measure of impairment, disability and handicap. It is intended to measure accurately general functional changes over the course of recovery and has found to be both valid and reliable.
  Scores range from 0 (normal) and 29 (extreme vegetative state).
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group Baseline | Treatment Group Baseline
Number analyzed (Participants) | 6 | 8
units on a scale | 1 (1.3) | 1.4 (1.1)

12. Secondary Outcome: Disability Rating Scale (DRS)
Description: as for outcome 11
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group 12 Weeks | Treatment Group 12 Weeks
Number analyzed (Participants) | 6 | 8
units on a scale | 0.7 (1) | 0.6 (0.3)

13. Secondary Outcome: Mini Mental Status Exam (MMSE)
Description: This outcome measure assess the participants Cognitive status. Scores range from 0 ( significantly impaired) -30 ( normal).
  A score of 23 or lower is indicative of cognitive impairment. In this study the score was used as a continuous variable.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group Baseline | Treatment Group Baseline
Number analyzed (Participants) | 6 | 8
units on a scale | 28.3 (1.6) | 27.1 (1.03)

14. Secondary Outcome: Mini Mental Status Exam (MMSE)
Description: as for outcome 13
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Group 12 Weeks | Treatment Group 12 Weeks
Number analyzed (Participants) | 6 | 8
units on a scale | 29.7 (0.5) | 29.0 (0.6)

ADVERSE EVENTS:
Time Frame: Through study completion
Groups:
- Escitalopram: Escitalopram was started at 10 mg per day and increased to 20 mg if deemed clinically necessary, at week 4. No medication changes were made after week.
Arm/Group | Placebo | Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No